CLINICAL TRIAL: NCT03970655
Title: Does the Addition of Epinephrine to Bilateral Ultrasound Guided Pterygopalatine Ganglion Block Reduce Bleeding During Functional Endoscopic Sinus Surgery (FESS)? A Pilot Study
Brief Title: Functional Endoscopic Sinus Surgery Study
Acronym: FESS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB201900782; OCR21462 (Other: UF OnCore)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Bupivacaine; Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): a single injection into the LEFT pterygopalatine fossa of 4 milliliters of 0.5% Bupivacaine or Ropivacaine with epinephrine 1:200.000 with the addition of 4 milligrams of dexamethasone (1ml) and a single injection into the RIGHT pterygopalatine fossa fo 4 milliliters of 0.5% Bupivacaine or Ropivacaine without epinephrine with the addition of 4 milligrams of dexamethasone (1mL) after the induction of general anesthesia. (total volume 5 ml per side)
  Interventions: Drug: Bupivacaine or Ropivacaine with epinephrine plus dexamethasone - Group 1
- Group 2 (Experimental): a single injection into the LEFT pterygopalatine fossa of 4 milliliters of 0.5% Bupivacaine or Ropivacaine without epinephrine with the addition of 4 milligrams of dexamethasone (1ml) and a single injection into the RIGHT pterygopalatine fossa of 4 milliliters of 0.5% Bupivacaine or Ropivacaine with epinephrine 1:200.00 with the addition of 4 milligrams of dexamethasone (1mL) after the induction of general anesthesia. (total volume 5 ml per side).
  Interventions: Drug: Bupivacaine or Ropivacaine with epinephrine plus dexamethasone - Group 2

INTERVENTIONS:
Drug: Bupivacaine or Ropivacaine with epinephrine plus dexamethasone - Group 1 — Group 1 will receive 4 ml of 0.5% Bupivacaine or Ropivacaine with epinephrine in the LEFT pterygopalatine fossa
  Arms: Group 1
Drug: Bupivacaine or Ropivacaine with epinephrine plus dexamethasone - Group 2 — Group 2 will receive 4 ml of 0.5% Bupivacaine or Ropivacaine with epinephrine in the RIGHT pterygopalatine fossa
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the effect of the addition of epinephrine to bilateral real time ultrasound guided pterygopalatine ganglion blocks on intra-operative bleeding and blood loss during functional endoscopic sinus surgery (FESS).

DETAILED DESCRIPTION:
FESS is the treatment of choice in patients with medically refractory chronic rhinosinusitis and chronic polypous rhinosinusitis. This surgery relies on minimal surgical site bleeding to be performed efficiently and safely. Hemorrhage during FESS decreases visibility of the surgical field and this increases the risk of vascular, orbital and intracranial complications as well as procedural failure. Thus the importance of minimizing surgical bleeding in this procedure. The maxillary artery is the primary blood supply for the sinuses and midface. Conceptually the application of epinephrine into the pterygopalatine fossa onto the maxillary artery with the block should result in constriction of this artery and subsequently, less bleeding from the surgical site. This randomized, double-blinded, controlled pilot study will investigate the utility of addition of epinephrine to bilateral pterygopalatine ganglion blocks performed under ultrasound guidance in minimizing surgical site bleeding and overall blood loss and the potential for shortening the surgical time.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting for bilateral FESS
2. Adult patients (>18 and < 90 years old)
3. Patient consents to participate
4. No underlying chronic pain condition
5. No underlying bleeding diathesis

Exclusion Criteria:

1. Patient refuses to consent
2. Patient requires revision or unilateral surgery
3. Patient requires surgery in addition to FESS
4. Age younger than 18 or older than 90 years
5. Any underlying chronic pain condition
6. History of bleeding diathesis
7. Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for block placement.
8. Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for research participation.
9. Vulnerable patient population

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
Change in Endoscopic Grading of Nasal Bleeding | Every 10 minutes up to 36 hours
  Endoscopic Grading of Nasal Bleeding will be calculated using the 0-5 point Boezaart surgical field grading scale; 0 being no bleeding and 5 being severe bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R Smith, Principal Investigator — University of Florida
Locations (1):
- UF Health of University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No